CLINICAL TRIAL: NCT00002035
Title: Double-Blind Comparison of the Efficacy of Continued Zidovudine Versus 2',3'-Dideoxyinosine (ddI) (BMY-40900) for the Treatment of Patients With AIDS or AIDS-Related Complex and Increasing Symptomatology Despite Treatment With Zidovudine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 039B; AI454-010
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: HIV Infections
Keywords: Didanosine; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To compare the efficacy and safety of orally administered didanosine (ddI) with orally administered zidovudine (AZT) in the treatment of patients who exhibit increasing clinical deterioration despite treatment with AZT.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed for Hematologic toxicity:

* Erythropoietin.
* Colony-Stimulating Factors.
* Allowed for prophylaxis of Pneumocystis carinii pneumonia (PCP):
* Aerosolized pentamidine.
* Trimethoprim/sulfamethoxazole.
* Dapsone.
* NOTE:
* If intravenous pentamidine is required for treatment of PCP, study drug should be suspended until one week after completion of intravenous pentamidine.
* Allowed:
* Prophylactic or suppressive therapy begun prior to study entry with the exception of neurotoxic agents (as defined in the protocol).

Concurrent Treatment:

Allowed:

* Transfusions for hematologic toxicity.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Active acute AIDS defining infection.
* Clinical evidence of acute pancreatitis in the last two years or chronic pancreatitis.
* Dementia of such severity that patient cannot give informed consent.
* Grade 2 or worse peripheral neuropathy as defined by Targeted Neuropathy Score (Schaumberg).
* Prior Cytomegalovirus disease requiring ongoing systemic ganciclovir therapy.
* Extensive Kaposi's sarcoma or other malignancy requiring systemic cytotoxic myelosuppressive or neurotoxic chemotherapy.
* Cardiomyopathy or the need for antiarrhythmic therapy.
* Inability to tolerate at least 600 mg per day of zidovudine (AZT).
* Seizures within the last 6 months or the need for anticonvulsant therapy.

Concurrent Medication:

Excluded:

* Ganciclovir (DHPG).
* Myelosuppressive or neurotoxic chemotherapy.
* Antiarrhythmic therapy.
* Anticonvulsant therapy.
* Neurotoxic agents (as defined in the protocol).
* NOTE:
* If intravenous pentamidine is required for treatment of Pneumocystis carinii pneumonia (PCP), study drug should be suspended until 1 week after completion of intravenous pentamidine.

Patients with the following are excluded:

* Symptoms and conditions defined in the Patient Exclusion Co-Existing Conditions field.
* Average of two sequential CD4 counts from SciCor Clinical Laboratories in the 30 days prior to study entry > 300 cells/mm3.

Prior Medication:

Excluded, participation in studies using:

* Dideoxyinosine (ddI).
* 2',3'-Dideoxy-2',3'-didehydrothymidine (d4T).
* Dideoxycytidine (ddC).
* Excluded within one month of study entry:
* Any other experimental antiretroviral compounds.

Patients must:

* Have documented HIV positivity via ELISA.
* Meet CDC criteria for AIDS or AIDS related complex (ARC).
* Have received zidovudine (AZT) for = or > 6 months and tolerated a dose of at least 500 mg per day without significant hematologic toxicity.
* Have no acute AIDS defining opportunistic infection, but may be receiving suppressive therapy for such infections.
* Demonstrate at least one of the following criteria for clinical deterioration despite AZT therapy within 4 weeks prior to study entry (8 weeks prior for weight loss):
* involuntary weight loss of more than 5 percent of the body weight occurring over the 8 week period prior to study entry, Karnofsky score = or > 50 but demonstrating a fall = or > 20 from previous level of functioning (assessment must be persistent on two occasions at least 14 days apart), unexplained fever of = or > 38 degrees C (despite evaluation defined in protocol) for more than 7 days, appearance of newly diagnosed oral hairy leukoplakia or oral candidiasis, or recurrence of a previously quiescent multidermatomal varicella-zoster, appearance of dermatologic afflictions (e.g. psoriasis, molluscum contagiosum, or newly diagnosed seborrheic dermatitis), appearance of chronic herpetic ulcers not responsive to acyclovir therapy.

Required:

* Zidovudine (AZT) for = or > 6 months prior to study entry.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Study Completion 1992-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- United States (17):
  - Univ of Arizona / Health Science Ctr, Tucson, Arizona
  - Yale Univ Med School, New Haven, Connecticut
  - G E Morey Jr, Fort Lauderdale, Florida
  - VP Med Services / HHCS Research Institute Inc, Orlando, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Edward Hines Veterans Administration Hosp, Hines, Illinois
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Harper Hosp, Detroit, Michigan
  - Albany Med College / AIDS Treatment Ctr, Albany, New York
  - Med College of Ohio, Toledo, Ohio
  - Univ of Pennsylvania / HIV Clinic, Philadelphia, Pennsylvania
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Audie L Murphy Veterans Administration Hosp, San Antonio, Texas
  - Univ of Utah School of Medicine, Salt Lake City, Utah
  - Dr Stephen L Green, Hampton, Virginia
  - Milwaukee County Med Complex, Milwaukee, Wisconsin
- UPR School of Medicine, San Juan, Puerto Rico

REFERENCES:
- [Background] Ruedy N, et al. Results of long term follow-up of a double blind study of ddI vs continued AZT among individuals with CD4s 200-500/mm3. Int Conf AIDS. 1994 Aug 7-12;10(2):16 (abstract no 358B)